CLINICAL TRIAL: NCT01218477
Title: Dasatinib (BMS-354825) Combined With SMO Inhibitor (BMS-833923; XL139) in CML With Resistance or Suboptimal Response to a Prior TKI
Brief Title: Dasatinib Combination Therapy With the Smoothened (SMO) Inhibitor BMS-833923 in Chronic Myeloid Leukemia (CML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-323; 2010-019480-11 (EudraCT Number)
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: Leukemia; (Chronic Myeloid Leukemia-Chronic Phase and Advanced)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; BMS-833923

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dasatinib, 100/140 mg QD (Experimental): Participants received dasatinib, 100/140 mg once daily (QD), depending on cohort (100 mg for those with chronic myeloid leukemia [CML]-chronic phase; 140 mg for those with CML-advanced phase)
  Interventions: Drug: Dasatinib
- Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD (Experimental): Participants received dasatinib, 100/140 mg once daily (QD), depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase) plus BMS-833923, 50 mg, QD
  Interventions: Drug: Dasatinib; Drug: BMS-833923
- Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID/QD (Experimental): Participants received BMS-833923, 100 mg twice daily (BID) for 7 days then once daily (QD) + dasatinib, 100/140 mg QD, depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
  Interventions: Drug: Dasatinib; Drug: BMS-833923
- Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD (Experimental): Participants received BMS-833923, 200 mg twice daily (BID) for 7 days then 200 mg once daily (QD) plus dasatinib, 100 /140 mg QD), depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
  Interventions: Drug: Dasatinib; Drug: BMS-833923

INTERVENTIONS:
Drug: Dasatinib — Oral tablets, 100-140 mg once daily, depending on cohort (100 mg for those with chronic myeloid leukemia [CML]-chronic phase; 140 mg for those with CML-advanced phase)
  Other Names: Sprycel
Drug: BMS-833923 — Oral capsules, 50-200 mg, depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
  Arms: Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD; Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID/QD; Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD

SUMMARY:
The purpose of the study is to determine the safety and tolerability of the combination of BMS-833923 plus dasatinib in patients with chronic myeloid leukemia.

ELIGIBILITY:
Key Inclusion Criteria

* Age ≥18 years
* Diagnosis of chronic myeloid leukemia (CML) and cytogenetic positive for the Philadelphia chromosome (Ph+), documented Ph+ cells on bone marrow assessment (BMA) ≤6 weeks prior to treatment
* Either chronic-phase CML, with <15% blasts in peripheral blood and bone marrow, or advanced-phase CML, including Ph+ acute lymphoblastic leukemia (ALL) (> 5% blasts) or hematologic progression with ≥15% blasts not in complete cytogenetic remission
* Resistance or suboptimal response to imatinib, dasatinib, or nilotinib and no known T315I/A Abl-kinase mutation.

Key Exclusion Criteria

* Known Abl-kinase T315I or T315A mutation
* CCyR at baseline
* Any serious or uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy
* Uncontrolled or significant cardiovascular disease
* Grade 3 or higher peripheral blood counts
* Serum calcium or phosphate below the lower limit of normal
* Baseline hypomagnesemia and amylase or lipase at least Grade 1 or higher
* Reduced renal function, defined as serum creatinine level >3*upper limit of normal
* Prior therapies for CML or Ph+ ALL permitted, with the following restriction:

  * Therapy permitted with corticosteroids, hydroxyurea, or anagrelide prior to starting treatment and during the first 4 weeks on study
  * 6 months or longer after stem cell transplantation
  * 28 days or longer after any investigational agent
  * 7 days or longer after any standard chemotherapy agent
  * Concomitant use of medications with a known risk of causing Torsades de Pointes
  * Concomitant use of strong inhibitors of the CYP3A4 isoenzyme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (3):
  - University Of California Medical Center, San Francisco, California
  - Sidney Kimmel Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Ut M.D. Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Local Institution, Hamilton, Ontario
  - Local Institution, Toronto, Ontario
- Local Institution, Helsinki, Finland
- France (2):
  - Local Institution, Bordeaux
  - Local Institution, Poitiers
- Local Institution, Frankfurt am Main, Germany
- Italy (2):
  - Local Institution, Bologna
  - Local Institution, Orbassano(To)
- Local Institution, Glasgow, United Kingdom

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 participants were enrolled; 27 were treated.
Groups:
- Dasatinib, 100/140 mg QD: Participants received dasatinib, 100/140 mg once daily (QD), depending on cohort cohort (100 mg for those with chronic myeloid leukemia [CML]-chronic phase; 140 mg for those with CML-advanced phase)
- Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD: Participants received dasatinib, 100/140 mg once daily (QD), depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase) plus BMS-833923, 50 mg QD
- Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID/QD: Participants received BMS-833923, 100 mg twice daily (BID), for 7 days then once daily (QD) + dasatinib, 100/140 mg QD, depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
- Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD: Participants received BMS-833923, 200 mg twice daily (BID) for 7 days then 200 mg once daily (QD) plus dasatinib, 100 /140 mg QD, depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
Period: Overall Study
Arm/Group | Dasatinib, 100/140 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID/QD | Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD
Started | 3 (Participants who received treatment) | 8 (Participants who received treatment) | 14 (Participants who received treatment) | 2 (Participants who received treatment)
Completed | 0 (Still receiving study drug) | 0 (Still receiving study drug) | 0 (Still receiving study drug) | 0 (Still receiving study drug)
Not Completed | 3 | 8 | 14 | 2
Not completed — Disease progression | 2 | 3 | 6 | 2
Not completed — Study drug toxicity | 0 | 2 | 5 | 0
Not completed — No longer meets study criteria | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Prepared for cell transplantation | 0 | 1 | 1 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 1 | 0
Not completed — Maximum clinical benefit | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study medication
Groups:
- Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD: Participants received dasatinib, 100/140 mg once daily (QD), plus BMS-833923, 50 mg, QD), depending on cohort cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
- Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD: Participants received BMS-833923, 200 mg twice daily (BID) for 7 days then once daily (QD) plus dasatinib, 100 /140 mg QD, depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
- Total: Total of all reporting groups
Arm/Group | Dasatinib, 100/140 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID/QD | Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD | Total
Number analyzed (Participants) | 3 | 8 | 14 | 2 | 27
Age, Continuous [Median (Full Range); unit: Years] | 43.0 [26.0 to 50.0] | 57.5 [36.0 to 68.0] | 55.5 [25.0 to 74.0] | 64.5 [56.0 to 73.0] | 56.0 [25.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7 | 1 | 15
  Male | 2 | 2 | 7 | 1 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1 | 7 | 11 | 2 | 21
  Black/African American | 1 | 1 | 2 | 0 | 4
  Other | 1 | 0 | 1 | 0 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Physicians use the ECOG scales and criteria to help determine the progression of a patient's disease, the disease's affect on the patient's daily living abilities, and appropriate treatment and prognosis. The scale runs from 0 (normal health) to 5 (death). Higher score=greater impairment. ECOG status scores: 0=fully active; 1=unable to perform strenuous activities, but light activity possible; 2=able to walk and manage self-care, but confined to a bed or chair <50% of the day; 3=confined to a bed or chair >50% of the day, but not bedridden; 4=completely disabled, bedridden; 5=dead.
  Participants
    0 | 2 | 2 | 11 | 1 | 16
    1 | 0 | 6 | 3 | 1 | 10
    2 | 1 | 0 | 0 | 0 | 1
Current leukemia diagnosis [Number; unit: Participants] — CML=chronic myeloid leukemia; ALL=acute lymphoblastic leukemia; Ph+=Philadelphia chromosome positive; Ph+ ALL=Philadelphia chromosome positive-acute lymphoblastic leukemia
  Participants
    Accelerated phase Ph+ CML | 1 | 0 | 2 | 0 | 3
    Chronic phase Ph+ CML | 1 | 8 | 8 | 2 | 19
    Myeloid blast | 1 | 0 | 0 | 0 | 1
    Ph+ ALL | 0 | 0 | 4 | 0 | 4
Current disease phase [Number; unit: Participants]
  CML-advanced phase | 2 | 0 | 6 | 0 | 8
  CML-chronic phase | 1 | 8 | 8 | 2 | 19
Previous medication for chronic myeloid leukemia [Number; unit: Participants]
  Dasatinib | 0 | 6 | 4 | 1 | 11
  Imatinib | 1 | 1 | 5 | 0 | 7
  Nilotinib | 2 | 1 | 5 | 1 | 9
Primary reason for eligibility [Number; unit: Participants]
  Cytogenetic progression | 1 | 1 | 4 | 0 | 6
  Hematologic progression | 1 | 1 | 4 | 1 | 7
  Suboptimal response | 1 | 6 | 6 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of BMS-833923 Plus Dasatinib in Chronic Myeloid Leukemia-Chronic Phase
Description: The following drug-related adverse events (AEs) occurring in the first 28 days of treatment were considered dose-limiting toxicities (DLT): Grade 4 hematologic AE lasting >7 days; ≥Grade 3 nonhematologic AE, despite medical intervention; ≥Grade 2 AE uncontrolled by medical intervention and requiring treatment interruption for >7 days. RP2D was that dose at which ≤1 of 6 patients had a DLT in the first 4 weeks of treatment. If <3 patients were DLT-evaluable, up to 6 additional patients entered the same dose level. Accrual to a dose level closed if 6 patients were enrolled and <3 were DLT-evaluable. If ≥3 patients at a dose level had no DLTs when a new patient enrolled, the dose was escalated to next level. If 1 DLT was observed in <6 patients, ≥6 patients were required; if no additional DLT was observed, the dose was escalated to the next highest level. If ≥2 DLTs were observed in <6 patients, that level exceeded the RP2D, and the dose was deescalated to the next lowest level.
Time Frame: Day 1 to Week 80, with observation for DLT in Weeks 5-8
Population: Participants who were dose-limiting toxicity (DLT)-evaluable (DLT-evaluable=received combination therapy on >21 of 28 days in Weeks 5 through 8 or interrupted treatment for drug-related AEs)
Measure: Number; unit: mg
Groups:
- Dasatinib, 100/140 mg QD, Plus BMS-833923, 50-200 BID/QD: Participants received BMS-833923 + dasatinib at 1 of 4 dosing levels: Dasatinib, 100 mg/140 mg QD, depending on cohort (100 mg for those with chronic myeloid leukemia [CML]-chronic phase; 140 mg for those with CML-advanced phase); BMS-833923, 50 mg once daily (QD) + dasatinib, 100 mg/140 mg QD; BMS-833923, 100 mg twice daily (BID) for 7 days, then 100 mg QD + dasatinib 100 mg/140 mg QD; or BMS-833923, 200 mg BID for 7 days, then 200 mg QD + dasatinib 100 mg/140 mg QD
Arm/Group | Dasatinib, 100/140 mg QD, Plus BMS-833923, 50-200 BID/QD
Number analyzed (Participants) | 24
mg | 50

2. Secondary Outcome: Percentage of Participants With a Major Cytogenetic Response (MCyR) in Chronic Myeloid Leukemia-Advanced Phase (CML-Adv) and Chronic Myeloid Leukemia-Chronic Phase (CML-CP)
Description: Cytogenetic response (CyR) was based on the proportion of Philadelphia chromosome-positive (Ph+) cells in metaphase analysis of bone marrow. Complete cytogenetic response (CCyR)=0 Ph+ cells; Partial CyR (PCyR)=1 to 35 Ph+ cells; Minor CyCR= 36-65 Ph+ cells; Minimal CyCR= 66-95 Ph+ cells; No response= >96 Ph+ cells. MCyR=CCyR + PCyR. Nilo=nilotinib; SOR=suboptimal response.
Time Frame: Day 1 to Week 80
Population: All patients without CCyR at dosing start date who received at least 4 weeks of dasatinib and had at least 1 on-treatment cytogenetic evaluation of the bone marrow data after at least 4 weeks on treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dasatinib, 100/140 mg QD, Plus BMS-833923, 50-200 BID/QD
Number analyzed (Participants) | 19
Percentage of participants
  CML-CP with imatinib or nilo resistance/SOR (n=6) | 66.7 [22.28 to 95.67]
  CML-CP with dasatinib resistance/SOR (n=10) | 20 [2.52 to 55.61]
  CML-Adv with imatinib or nilo resistance/SOR (n=3) | 66.7 [9.43 to 99.16]

3. Secondary Outcome: Percentage of Participants With a Major Hematologic Response (MHR) in Chronic Myeloid Leukemia-Advanced Phase (CML-Adv) and Chronic Myeloid Leukemia-Chronic Phase (CML-CP)
Description: MHR was defined as complete hematologic response (CHR) or no evidence of leukemia (NEL). CHR for CML-Adv criteria: white blood cell count (WBC) ≤upper limit normal; absolute neutrophil count (ANC) ≥1,000/mm^3; platelets ≥100,000/mm^3; no blasts or promyelocytes in peripheral blood (PB); basophils <5% in PB; myelocytes + metamyelocytes < 5% in PB; no extramedullary involvement; blasts must be <5%, if bone marrow assessment (BMA) performed. NEL had same criteria, but with lower thresholds for reconstitution of PB counts, as follows: Platelets ≥ 20,000/mm^3 or ANC >500/mm^3. Confirmed MHR obtained if these criteria met and maintained for ≥28 days. CHR for CML-CP criteria WBC ≤10,000/mm^3; platelets <450,000/mm^3; basophils <5% in PB; no blasts or promyelocytes in PB; myelocytes + metamyelocytes <5% in PB; no extramedullary involvement; blasts must be <5% if BMA performed. Confirmed CHR obtained if these criteria met and maintained for ≥28 days. Nilo=nilotinib; SOR=suboptimal response.
Time Frame: Day 1 to Week 80
Population: Patients without complete hematologic response at dosing start date who received at least 4 weeks of dasatinib and who had at least 1 on-treatment evaluation of both peripheral blood counts and bone marrow cytogenetic response after at least 4 weeks on treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dasatinib, 100/140 mg QD, Plus BMS-833923, 50-200 BID/QD
Number analyzed (Participants) | 8
Percentage of participants
  CML-CP with imatinib or nilo resistance/SOR (n=2) | 50 [1.26 to 98.74]
  CML-CP with dasatinib resistance/SOR (n=5) | 60 [14.66 to 94.73]
  CML-CP with imatinib or nilo resistance/SOR (n=1) | 100 [2.5 to 100]

4. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, Adverse Events (AEs) Leading to Discontinuation, Drug-related AEs Leading to Discontinuation, at Least 1 Drug-related AE, and Dose-limiting Toxicities
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment and may or may not be related to treatment. SAE=an untoward medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=having certain, probable, possible, or missing relationship to study drug. The following drug-related AEs occurring during the first 28 days of treatment with both agents were considered to be dose-limiting toxicities (DLTs): Grade 4 hematologic AE lasting >7 days; ≥Grade 3 nonhematologic AE, despite adequate medical intervention; ≥Grade 2 AE not controlled by medical intervention and requiring treatment interruption for >7 days.
Time Frame: Day 1 to Week 80, continuously, with observation for dose-limiting toxicities (DLTs) in Weeks 5-8
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Groups:
- Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD: Participants received BMS-833923, 200 mg twice daily (BID) for 7 days, then once daily (QD), plus dasatinib, 100 /140 mg QD, depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
Arm/Group | Dasatinib, 100/140 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID/QD | Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD
Number analyzed (Participants) | 3 | 8 | 14 | 2
Participants
  Death | 1 | 0 | 2 | 0
  SAEs | 1 | 3 | 5 | 0
  Drug-related SAEs | 0 | 1 | 0 | 0
  AEs leading to discontinuation | 1 | 2 | 5 | 0
  Drug-related AEs leading to discontinuation | 0 | 2 | 5 | 0
  At least 1 drug-related AE | 0 | 8 | 13 | 2
  DLTs | NA — DLTs were only defined for treatment with both dasatinib and BMS-833923 | 0 | 2 | 1

5. Secondary Outcome: Number of Participants With Grade 3-4 Abnormalities on Laboratory Test Results
Description: ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; ULN=upper limit of normal. Abnormalities were graded according to the Common Toxicity Criteria of the National Cancer Institute from 1 (least severe) to 4 (life threatening). ANC (*10^9): Grade 3, <1.0- 0.5; Grade 4, <0.5. Hemoglobin (mmol/L): Grade 3, <4.9-4.0; Grade 4, <4.0. Platelet count (*10^9/L): Grade 3, <50.0-25.0; Grade 4, <25. WBCs (*10^9): Grade 3, <2.0-1.0; Grade 4, <1.0. Hypocalcemia (mmol/L): Grade 3, <1.75-1.5; Grade 4, <1.5. Hyperkalemia (mmol/L): Grade 3, >6.0-7.0; Grade 4, >7.0. Hypokalemia (mmol/L): Grade 3, <3.0-2.5; Grade 4, <2.5. Hyponatremia (mmol/L), Grade 3, <130-120; Grade 4, <120. Hypermagnesemia (mg/dL): Grade 3, >1.23-3.30; Grade 4, >3.30. Phosphorus (mmol/L): Grade 3, <0.6-0.3; Grade 4, <0.3. Lipase (*ULN): Grade 3, >2.0-5.0; Grade 4, >5.0.
Time Frame: Day 1 to Week 80
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Groups:
- Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD: Participants received dasatinib, 100/140 mg once daily (QD), depending on cohort cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase) plus BMS-833923, 50 mg, QD
- Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID: Participants received BMS-833923, 100 mg twice daily (BID), for 7 days, followed by dasatinib, 100/140 mg once daily (QD)
Arm/Group | Dasatinib, 100/140 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 50 mg QD | Dasatinib, 100/140 mg QD + BMS-833923, 100 mg BID | Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD
Number analyzed (Participants) | 3 | 8 | 14 | 2
Participants
  Absolute neutrophil count (ANC) | 0 | 0 | 5 | 0
  Hemoglobin | 0 | 0 | 3 | 0
  Platelet count (n=1, 8, 14, 2) | 1 | 0 | 3 | 0
  White blood cell count (WBC) | 0 | 0 | 3 | 0
  Hypocalcemia | 0 | 0 | 1 | 0
  Hyperkalemia | 0 | 1 | 0 | 0
  Hypokalemia | 0 | 0 | 2 | 0
  Hyponatremia | 0 | 1 | 0 | 0
  Hypermagnesemia | 0 | 0 | 1 | 0
  Phosphorus, inorganic (n=3, 8, 12, 2) | 0 | 0 | 3 | 0
  Lipase, total (n=3, 3,14, 2) | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Groups:
- Dasatinib, 100/140 mg QD: Participants received dasatinib, 100/140 mg once daily (QD) (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
- Dasatanib, 100/140 mg QD + BMS-833923, 50 mg QD: Participants received dasatanib, 100/140 mg once daily (QD), as oral tablets plus BMS-833923, 50 mg, QD (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
- Dasatanib, 100/140 mg QD + BMS-833923, 100 mg BID/QD: Participants received BMS-833923, 100 mg twice daily (BID) for 7 days then once daily (QD) + dasatanib, 100/140 mg QD, depending on cohort (100 mg for those with CML-chronic phase; 140 mg for those with CML-advanced phase)
Arm/Group | Dasatinib, 100/140 mg QD | Dasatanib, 100/140 mg QD + BMS-833923, 50 mg QD | Dasatanib, 100/140 mg QD + BMS-833923, 100 mg BID/QD | Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/8 | 5/14 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 8/8 | 14/14 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100/140 mg QD (N=3) | Dasatanib, 100/140 mg QD + BMS-833923, 50 mg QD (N=8) | Dasatanib, 100/140 mg QD + BMS-833923, 100 mg BID/QD (N=14) | Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD (N=2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Uterine carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100/140 mg QD (N=3) | Dasatanib, 100/140 mg QD + BMS-833923, 50 mg QD (N=8) | Dasatanib, 100/140 mg QD + BMS-833923, 100 mg BID/QD (N=14) | Dasatinib, 100 /140 mg QD+ BMS-833923, 200 mg BID/QD (N=2)
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Amylase (Investigations) | 0 | 2 | 0 | 0
Amylase increased (Investigations) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 5 | 10 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 3 | 7 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Blood creatinine (Investigations) | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 7 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 0
Lipase (Investigations) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 4 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Herpes dermatitis (Infections and infestations) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 8 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0
Asthenia (General disorders) | 0 | 1 | 2 | 0
Blood cholesterol (Investigations) | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 2 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 11 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 3 | 4 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Bristol-Myers Squibb discontinued research in the area of smoothened inhibitors. This study was completed early and limited efficacy data was published in a synoptic clinical study report .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.